CLINICAL TRIAL: NCT03275870
Title: Pilot Study of Hydroxychloroquine for the Treatment of Hidradenitis Suppurativa
Brief Title: Hydroxychloroquine for the Treatment of Hidradenitis Suppurativa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elena Gonzalez Brant, MD (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Elena Gonzalez Brant, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050057
Record Dates: First submitted 2017-08-31; First posted 2017-09-08 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Hidradenitis Suppurativa; Hidradenitis; Acne Inversa; Boils; Follicular Occlusion Triad; Follicular Occlusion Tetrad
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Furunculosis | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hydroxychloroquine treatment (Experimental): Hydroxychloroquine 200mg BID for 6 months
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Treatment of patients with hidradenitis suppurativa with hydroxychloroquine 200mg BID for 6 months
  Other Names: Plaquenil

SUMMARY:
Hidradenitis suppurativa (HS) is an under-recognized and debilitating disease. Patients suffer from recurring painful abscesses and scarring in their armpits, under the breasts, groin and other areas of the body. The cause of the disease is still unknown and common treatments are only sometimes effective. Overactivity of the immune system has been associated with HS and molecules that cause inflammation have been found in the skin from people with HS. Current therapies have long-term risks including antibiotic resistance and the investigators aim to find new safe and effective therapies for HS.

Hydroxychloroquine is a medication that has been used safely in other diseases for many years. The investigators believe that hydroxychloroquine has the potential to improve HS through multiple mechanisms. Patients enrolled in this study will be treated with hydroxychloroquine for 6 months. The investigators also aim to look at the blood of patients with HS to look for inflammatory molecules that we could possibly target for the treatment of HS. Blood samples will be taken at baseline and following 6 months of treatment.

DETAILED DESCRIPTION:
Hidradenitis suppurativa is a debilitating and mutilating disease and its pathogenesis is still poorly understood. It involves the development of recurrent, painful nodules in intertriginous areas that become inflamed, form abscesses that may rupture, and develop chronic fistula tracts. The cause of hidradenitis suppurativa (HS) is thought to be multifactorial and may begin with follicular occlusion and rupture, leading to a cascade of inflammatory responses in susceptible individuals. The disease has been associated with high body mass index, smoking and genetic predisposition. There is a known association between HS and the metabolic syndrome, an association that remains after controlling for body mass index. HS predominantly affects women and ethnic minorities and the prevalence is thought to be as high as 2%, although embarrassment and lack of awareness may lead to an underestimate of the true burden of disease.

Although HS is a fairly common disease, relatively little is understood about its pathogenesis. Immune dysregulation is thought to play a role in disease development. Increased levels of interleukin (IL)-12, IL-17, IL-23, tumor necrosis factor α, IL-10 and IL-1β were found to be expressed in lesional skin of HS patients. Recent studies have also identified elevated levels of IL-17 in the serum of patients with HS.

HS is associated with a significant impact on patient quality of life. Patients suffer from both the physical and psychological impact of disease. Many therapies have been used to treat HS, from topical antibiotics to oral retinoids to radical surgeries, but all have limited efficacy. Despite efforts to control disease, many patients live with chronic wounds and disability. The decision about appropriate therapy for HS, especially in the early stages, is mainly based on expert opinion, anecdotal evidence, and small studies. Topical and systemic antimicrobial treatments are often used as first line therapies, although studies have repeatedly shown that the abscesses of HS are sterile or contain only normal flora. The mechanism of improvement with antimicrobials may be through alterations in the local microbiome. Significant improvement in disease has been seen with dual therapy with twice daily use of 300mg rifampicin and 300mg clindamycin, neither of which have an FDA indication for use in HS. Doxycycline is used frequently in HS, but little evidence supports this. Despite success with the above therapies, the risk of antimicrobial resistance is real, and is increased with frequent and prolonged use of these medications in HS. Teratogenic effects, gastrointestinal upset, and photosensitivity with use of tetracyclines, risk for clostridium difficile colitis with clindamycin, and antimicrobial resistance with rifampicin highlight a need for safer and effective therapeutic options for the treatment of early HS.

For more advanced disease (Hurley stage II and III), the tumor necrosis factor inhibitor adalimumab is the only FDA approved biologic treatment for HS. It has shown promise in severe disease, but only ~50% of patients achieved a clinical response at 12 weeks, and this clinical response declined over time. Additionally, newer biologic therapies have been used in small numbers of patients with HS with variable results. Importantly, the cost of these medications is considerable.

Hydroxychloroquine, initially developed as an antimalarial, has been used successfully for over 70 years in the treatment of autoimmune disease. Its mechanism of action is still poorly understood, but it has been shown to have many varied immunomodulatory properties. Evidence suggests that hydroxychloroquine has an effect on inflammatory disease through decreasing levels of TNFα and Th-17 cytokines (including IL-6, IL-17, and IL-22). Additionally, studies have shown a beneficial effect of hydroxychloroquine on lipid metabolism and glucose. Patients with rheumatoid arthritis (which similarly to HS has an independent association with cardiovascular disease) who were treated with hydroxychloroquine had an overall decreased incidence of cardiovascular events. Hydroxychloroquine has a relatively benign safety profile, with retinopathy being the most concerning long term side effect. The retinopathy caused by hydroxychloroquine is reversible if identified early, and standard protocols for the use of this medication include yearly ophthalmologic examination.

Patients with HS suffer daily from the physical and psychological effects of their disease. Despite insufficient data about disease progression and prognosis, early intervention with safe and effective therapies is our goal. Hydroxychloroquine has never been used to treat HS, but the good safety profile, based on many years of usage in other autoimmune diseases, and known ability to modify many of the aberrant metabolic and inflammatory components of HS make it an ideal candidate therapy for this debilitating disease.

Research activities:

1. Treatment with hydroxychloroquine 200mg twice daily. Treatment length will be 6 months. Patients will be allowed to continue or initiate use of topical therapies during the study.
2. Telephone call to assess toxicity after 1 month of treatment
3. Assessment of hidradenitis suppurativa disease activity using Sartorius scoring at baseline, and after 3 and 6 months of treatment
4. Collection of patient serum at baseline and after 6 months of treatment
5. Quality of life questionnaire at baseline, 3 and 6 months
6. Follow up telephone call at ~9 and 12 months (3 and 6 months after therapy completion) to assess for toxicity
7. Baseline ophthalmologic exam for patients on hydroxychloroquine will be conducted within the first year of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with hidradenitis suppurativa Hurley stage I or II

Exclusion Criteria:

* Current systemic immunosuppression, current use of biologic medication or use of these medications in the prior 3 months, patients with known retinal disease, hepatic disease (HCV, cirrhosis, aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of normal), psoriasis, porphyria cutanea tarda, platelets < 50,000/ul, leukocytes <4000/ul, or Hb<8g/dl), pregnant patients or women trying to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena M Gonzalez Brant, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gonzalez-Lopez MA, Hernandez JL, Lacalle M, Mata C, Lopez-Escobar M, Lopez-Mejias R, Portilla V, Fuentevilla P, Corrales A, Gonzalez-Vela MC, Gonzalez-Gay MA, Blanco R. Increased prevalence of subclinical atherosclerosis in patients with hidradenitis suppurativa (HS). J Am Acad Dermatol. 2016 Aug;75(2):329-35. doi: 10.1016/j.jaad.2016.03.025. Epub 2016 Jun 8. PMID 27287248
- [Background] Nicola WG, Khayria MI, Osfor MM. Plasma testosterone level and the male genital system after chloroquine therapy. Boll Chim Farm. 1997 Jan;136(1):39-43. PMID 9080720
- [Background] Garg A, Lavian J, Lin G, Strunk A, Alloo A. Incidence of hidradenitis suppurativa in the United States: A sex- and age-adjusted population analysis. J Am Acad Dermatol. 2017 Jul;77(1):118-122. doi: 10.1016/j.jaad.2017.02.005. Epub 2017 Mar 9. PMID 28285782
- [Background] Schlapbach C, Hanni T, Yawalkar N, Hunger RE. Expression of the IL-23/Th17 pathway in lesions of hidradenitis suppurativa. J Am Acad Dermatol. 2011 Oct;65(4):790-798. doi: 10.1016/j.jaad.2010.07.010. PMID 21641076
- [Background] van der Zee HH, de Ruiter L, van den Broecke DG, Dik WA, Laman JD, Prens EP. Elevated levels of tumour necrosis factor (TNF)-alpha, interleukin (IL)-1beta and IL-10 in hidradenitis suppurativa skin: a rationale for targeting TNF-alpha and IL-1beta. Br J Dermatol. 2011 Jun;164(6):1292-8. doi: 10.1111/j.1365-2133.2011.10254.x. Epub 2011 May 17. PMID 21332464
- [Background] Matusiak L, Szczech J, Bieniek A, Nowicka-Suszko D, Szepietowski JC. Increased interleukin (IL)-17 serum levels in patients with hidradenitis suppurativa: Implications for treatment with anti-IL-17 agents. J Am Acad Dermatol. 2017 Apr;76(4):670-675. doi: 10.1016/j.jaad.2016.10.042. Epub 2016 Dec 29. PMID 28041632
- [Background] von der Werth JM, Jemec GB. Morbidity in patients with hidradenitis suppurativa. Br J Dermatol. 2001 Apr;144(4):809-13. doi: 10.1046/j.1365-2133.2001.04137.x. PMID 11298541
- [Background] Andersen RK, Jemec GB. Treatments for hidradenitis suppurativa. Clin Dermatol. 2017 Mar-Apr;35(2):218-224. doi: 10.1016/j.clindermatol.2016.10.018. Epub 2016 Oct 27. PMID 28274363
- [Background] Fischer AH, Haskin A, Okoye GA. Patterns of antimicrobial resistance in lesions of hidradenitis suppurativa. J Am Acad Dermatol. 2017 Feb;76(2):309-313.e2. doi: 10.1016/j.jaad.2016.08.001. Epub 2016 Oct 11. PMID 27742173
- [Background] Kimball AB, Okun MM, Williams DA, Gottlieb AB, Papp KA, Zouboulis CC, Armstrong AW, Kerdel F, Gold MH, Forman SB, Korman NJ, Giamarellos-Bourboulis EJ, Crowley JJ, Lynde C, Reguiai Z, Prens EP, Alwawi E, Mostafa NM, Pinsky B, Sundaram M, Gu Y, Carlson DM, Jemec GB. Two Phase 3 Trials of Adalimumab for Hidradenitis Suppurativa. N Engl J Med. 2016 Aug 4;375(5):422-34. doi: 10.1056/NEJMoa1504370. PMID 27518661
- [Background] Rainsford KD, Parke AL, Clifford-Rashotte M, Kean WF. Therapy and pharmacological properties of hydroxychloroquine and chloroquine in treatment of systemic lupus erythematosus, rheumatoid arthritis and related diseases. Inflammopharmacology. 2015 Oct;23(5):231-69. doi: 10.1007/s10787-015-0239-y. Epub 2015 Aug 6. PMID 26246395
- [Background] van den Borne BE, Dijkmans BA, de Rooij HH, le Cessie S, Verweij CL. Chloroquine and hydroxychloroquine equally affect tumor necrosis factor-alpha, interleukin 6, and interferon-gamma production by peripheral blood mononuclear cells. J Rheumatol. 1997 Jan;24(1):55-60. PMID 9002011
- [Background] Silva JC, Mariz HA, Rocha LF Jr, Oliveira PS, Dantas AT, Duarte AL, Pitta Ida R, Galdino SL, Pitta MG. Hydroxychloroquine decreases Th17-related cytokines in systemic lupus erythematosus and rheumatoid arthritis patients. Clinics (Sao Paulo). 2013 Jun;68(6):766-71. doi: 10.6061/clinics/2013(06)07. PMID 23778483
- [Background] Hage MP, Al-Badri MR, Azar ST. A favorable effect of hydroxychloroquine on glucose and lipid metabolism beyond its anti-inflammatory role. Ther Adv Endocrinol Metab. 2014 Aug;5(4):77-85. doi: 10.1177/2042018814547204. PMID 25343023
- [Background] Sharma TS, Wasko MC, Tang X, Vedamurthy D, Yan X, Cote J, Bili A. Hydroxychloroquine Use Is Associated With Decreased Incident Cardiovascular Events in Rheumatoid Arthritis Patients. J Am Heart Assoc. 2016 Jan 4;5(1):e002867. doi: 10.1161/JAHA.115.002867. PMID 26727968

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine Treatment
Started | 17
Completed | 3
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxychloroquine Treatment
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 38.9 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  Black | 3
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Severity
Description: Comparison of baseline and post-treatment Sartorius severity scoring Sartorius scoring: minimum 0, no maximum, higher scores mean a worse outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydroxychloroquine Treatment
Number analyzed (Participants) | 3
score on a scale
  Baseline sartorius score | 23.3 (16.2)
  6 month sartorius score | 17.7 (14.4)
Statistical Analysis 1: Comparison: Hydroxychloroquine Treatment; Test type: Other; p = 0.042, t-test, 2 sided — p value <0.05 used as threshold for significance

2. Secondary Outcome: Change in Quality of Life
Description: Comparison of baseline and post-treatment self-reported quality of life Dermatology Life Quality Index score: minimum 0, maximum 30. higher scores mean worse outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydroxychloroquine Treatment
Number analyzed (Participants) | 3
score on a scale
  Baseline DLQI score | 14.7 (11)
  6 month DLQI score | 6 (7.9)
Statistical Analysis 1: Comparison: Hydroxychloroquine Treatment; Test type: Other; p = 0.213, t-test, 2 sided — P value of <0.05 used as threshold for significance

ADVERSE EVENTS:
Time Frame: 13 months
Description: Patients were periodically asked about side effects by a telephone call 1 month after starting treatment, at the 3 and 6 month follow up visit.
  They were evaluated for blurred vision, changes in vision, diarrhea, nausea, vomiting, headache, pruritus, anorexia and abdominal pain
Arm/Group | Hydroxychloroquine Treatment
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine Treatment (N=17)
Nausea (Gastrointestinal disorders) | 2 (2)
headache (Nervous system disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
We did not reach the target number of participants needed to achieve target power and statistically reliable results leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03275870/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03275870/Prot_SAP_003.pdf